CLINICAL TRIAL: NCT02998762
Title: CAN-BIND (Canadian Biomarker Integration Network for Depression): Long-Term Follow Up Study
Brief Title: Long-Term Follow Up Study
Acronym: CAN-BIND LTFU
Status: Completed | Type: Observational
Sponsor: Sidney Kennedy (Other)
Collaborators: Queen's University (Other); McMaster University (Other); University of Calgary (Other); University of British Columbia (Other)
Responsible Party: Sponsor-Investigator, Sidney Kennedy, Senior Scientist, Psychiatrist, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Other Study IDs: 15-9055-AE
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Major Depressive Disorder
Keywords: major depression; major depressive disorder; biomarkers; MDD; long term follow up
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The LTFU study will conduct a naturalistic follow up of the well characterized CAN-BIND study population of patients every six months and continuing over a five-year period. This will provide information on the longitudinal progress in mood, functioning, and quality of life of the CAN-BIND sample with a view towards long-term outcome and treatment.

DETAILED DESCRIPTION:
This is a long-term follow up study of the 'Canadian Biomarker Integration Network in Depression' (CAN-BIND) study. The CAN-BIND study examines biological markers of antidepressant treatment response. The examined biomarkers included clinical, imaging, and genetic components. The Long Term Follow up (LTFU) study will continue to follow the patients in this study each six months over a five year period. By doing so, a comprehensive clinical outcome data on a well characterized cohort of depressed patients will be obtained.

The research team will conduct a naturalistic study of CAN-BIND participants and will monitor the longitudinal progress in mood, functioning, and quality of life, with a view towards advising future treatment options. Each patient completing CAN-BIND will be asked to participate in the LTFU study.

ELIGIBILITY:
Inclusion Criteria:

* Each patient completing the 16 weeks of CAN-BIND who have previously met DSM-IV-TR criteria for Major Depressive Episode (MDE) in MDD as determined by MINI.

Exclusion Criteria:

* Any Axis I diagnosis, other than MDD, that is considered the primary diagnosis.
* Bipolar I or Bipolar II diagnosis (lifetime), MDD with psychotic features (lifetime), schizophrenia or schizoaffective disorder.
* Presence of a significant Axis II diagnosis (borderline, antisocial).
* High suicidal risk, defined by clinician judgement.
* History of drug or alcohol use, with a severity of at least moderate or severe, according to DSM criteria, within the previous 6 months.
* Presence of significant neurologic disorder, head trauma, or other unstable medical conditions.
* Subject has any condition, for which in the opinion of the investigator, participation would not be in the interest of the subject (e.g. compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Each patient completing the 16 weeks of CAN-BIND who have previously met DSM-IV-TR criteria for Major Depressive Episode (MDE) in MDD as determined by MINI.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) (Montgomery and Asberg 1979) scores from CAN-BIND baseline | Every six months up to Year 5
  Clinical response (equal to or greater than 50% reduction in MADRS scores from CAN-BIND baseline); Relapse is determined if the MADRS score is greater than or equal to 22 or there is suicidal ideation with intent, or suicidal behaviour.

SECONDARY OUTCOMES:
Longitudinal Interval Follow-up Evaluation (LIFE) (Keller et al., 1978) | Every six months up to Year 5
  The LIFE is a clinician-rated interview that provides a structure for collecting and coding data on the longitudinal course of psychopathology. It allows for precise dating of onset and offset of symptoms (including sub-syndromal symptoms) and ranks severity on a week by week basis.
Life Events and Difficulties Schedule (LEDS) (Brown & Harris, 1978) | Every six months up to Year 5
  The LEDS is a semi-structured interview that collects detailed contextual information regarding acute stressful life events and chronic difficulties in several domains.

OTHER OUTCOMES:
Quick Inventory Depressive Symptomatology-Self Report (QIDS-SR) (Rush et al., 2003) | Every six months up to Year 5
  The QIDS-SR is a 16 item scale used to assess the severity of depressive illness derived from the 30-item Inventory of Depressive Symptomatology (IDS). The scale includes questions on mood, sleep and level of interest, and takes 5-10 minutes to complete.
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) (Endicott et al., 1993) | Every six months up to Year 5
  This 16-item questionnaire contains questions about your general life satisfaction on aspects such as physical health, leisure time and overall sense of well-being. Each item is scored on a 5-point scale (very poor to very good); higher scores indicate greater satisfaction and enjoyment. It takes 5 minutes to complete.
Sheehan Disability Scale - Visual Analog Scale (SDS-VAS) (Sheehan et al., 1996) | Every six months up to Year 5
  The SDS-VAS is a self-rated questionnaire that assesses functional disability and impairment due to psychiatric symptoms. The SDS-VAS consists of three functional impairment items and two items related to productivity losses due to the symptoms and impairment. Impairment is evaluated with the 10-point self-rated social life and family life/home responsibilities subscales of the Sheehan Disability Scale (0, none; 1-3, mild; 4-6, moderate; 7-9, marked; 10, extreme). Significant impairment for each subscale was defined by a rating of 7 or higher.
The Dimensional Anhedonia Rating Scale (DARS) (Rizvi et al., 2015) | Every six months up to Year 5
  The DARS is a new measure of anhedonia developed to address the limitations of the existing scales. It extends the concept of anhedonia to assess desire, motivation, effort and consummatory pleasure across four domains: pastimes/hobbies, food/drink, social activities and sensory experiences. Individuals are asked to list their own examples within each domain and respond to standardized questions on a Likert scale according to how they are feeling "right now".
World Health Organization Quality of Life Short Version (WHOQOL-BREF) (Orley & Kuyken, 1994) | Every six months up to Year 5
  The WHOQOL-BREF is a 26-item self-rated questionnaire that assesses perceived quality of life across four domains. The domains of health assessed include physical health, psychological health, social relationships and environment. Domain scores and global scores can be generated. The questions are related to aspects of the patient's life in the last four weeks.
Brief Symptom Inventory (BSI-53) (Derogatis et al., 1993) | Every six months up to Year 5
  The BSI-53 is a 53-item self-rated questionnaire that assesses depression across nine symptom dimensions. The nine dimensions are somatization, obsession-compulsion, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism. The number and intensity of symptomatology is given by three indices, the Global Severity Index, Positive Symptom Distress Index and Positive Symptom Total (PST). Each item is ranked on a 5-point scale from 0 (not at all) to 4 (extremely), and rankings represent intensity of distress over the past week.
Generalized Anxiety Disorder 7-item (GAD-7) (Spitzer et al., 2006) | Every six months up to Year 5
  The GAD-7 is a 7-item self-rated questionnaire with good reliability and validity for assessing generalized anxiety disorder and its severity over the past two weeks. Items are ranked on a 4-point scale from 0 (not at all sure) to 3 (nearly every day), providing a total severity score from 0 to 21.
Pittsburgh Sleep Quality Index (PSQI) (Buysse at al., 1989) | Every six months up to Year 5
  The PSQI is a self-rated questionnaire specifically designed to measure sleep quality. The questionnaire includes questions on sleep duration, sleep disturbance, sleep latency, day dysfunction due to sleepiness, sleep efficiency, overall sleep quality and need for medication to sleep. This questionnaire takes less than 5 minutes to complete.
Copenhagen Burnout Inventory (CBI) (Kristensen et al., 2005) | Every six months up to Year 5
  The CBI consists of three scales measuring personal burnout, work-related burnout, and client-related burnout, for use in different domains. Each subscale on the CBI is scored from a range of 0 to 100. Respondents who gained an average score of 50 or higher on each of the scales are deemed to have a positive response to the screen and to warrant further investigation by a mental health professional.

CONTACTS AND LOCATIONS:
Overall Officials: Sidney H. Kennedy, MD, Principal Investigator — University Health Network, Toronto; Shane McInerney, MD, Principal Investigator — University Health Network, Toronto
Locations (5):
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
This study is funded in part by the Ontario Brain Institute (OBI). Data collected from this study is entered into a research database called "Brain-CODE", deployed at a High Performance Computer Virtual Lab (HPCVL). The HPCVL supports the regulatory-compliant (e.g., 21 CRF Part 11, HIPAA, PIPEDA) processes for securing privacy of healthcare data.

REFERENCES:
- [Background] Kennedy SH, Downar J, Evans KR, Feilotter H, Lam RW, MacQueen GM, Milev R, Parikh SV, Rotzinger S, Soares C. The Canadian Biomarker Integration Network in Depression (CAN-BIND): advances in response prediction. Curr Pharm Des. 2012;18(36):5976-89. doi: 10.2174/138161212803523635. PMID 22681173
- [Background] Vaccarino AL, Evans KR, Kalali AH, Kennedy SH, Engelhardt N, Frey BN, Greist JH, Kobak KA, Lam RW, MacQueen G, Milev R, Placenza FM, Ravindran AV, Sheehan DV, Sills T, Williams JB. The Depression Inventory Development Workgroup: A Collaborative, Empirically Driven Initiative to Develop a New Assessment Tool for Major Depressive Disorder. Innov Clin Neurosci. 2016 Oct 1;13(9-10):20-31. eCollection 2016 Sep-Oct. PMID 27974997
- [Background] Lam RW, Milev R, Rotzinger S, Andreazza AC, Blier P, Brenner C, Daskalakis ZJ, Dharsee M, Downar J, Evans KR, Farzan F, Foster JA, Frey BN, Geraci J, Giacobbe P, Feilotter HE, Hall GB, Harkness KL, Hassel S, Ismail Z, Leri F, Liotti M, MacQueen GM, McAndrews MP, Minuzzi L, Muller DJ, Parikh SV, Placenza FM, Quilty LC, Ravindran AV, Salomons TV, Soares CN, Strother SC, Turecki G, Vaccarino AL, Vila-Rodriguez F, Kennedy SH; CAN-BIND Investigator Team. Discovering biomarkers for antidepressant response: protocol from the Canadian biomarker integration network in depression (CAN-BIND) and clinical characteristics of the first patient cohort. BMC Psychiatry. 2016 Apr 16;16:105. doi: 10.1186/s12888-016-0785-x. PMID 27084692
- See also: CAN-BIND Study Website — http://www.canbind.ca